CLINICAL TRIAL: NCT05777811
Title: Effect of Different Recession Coverage Approaches on Sites With Shallow Vestibule Depth
Brief Title: The Relationship Between Root Coverage Procedures and Buccal Vestibular Depth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gencay Keceli, Assoc. Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Buccal Vestibule Depth
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Shallow Vestibular Depth; Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Patients were randomly assigned to either the Vertically Coronally Advanced Flap (n=25) group or the Free Gingival Graft (n=25) group by one of the authors, with an allocation ratio of 1:1, using a computer-generated program after the successful completion of Phase I periodontal treatment. One calibrated author applied the surgical technique and recorded all clinical variables. The surgeon opened the labeled envelope containing the intervention name.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vertically Coronally advanced flap combined with connective tissue graft (Active Comparator)
  Interventions: Procedure: Vertically coronally advanced flap combined with connective tissue graft.
- Free Gingival Graft (Active Comparator)
  Interventions: Procedure: Free gingival graft

INTERVENTIONS:
Procedure: Vertically coronally advanced flap combined with connective tissue graft. — The exposed root surfaces are planed with Gracey 1-2 curettes. An intrasulcular incision is made with a blade on the buccal aspects of the involved teeth. The incision is extended horizontally to the adjacent papilla. Then, slightly divergent vertical releasing incisions are carried 2 mm beyond the mucogingival junction. A full-thickness flap is raised with a periosteal elevator towards the mucogingival junction. After that, a partial-thickness dissection is carried out in the apical direction to release muscle tension and provide coronal advancement of the flap. The adjacent papillae are de-epithelialized. The connective tissue graft (CTG) is harvested from the lateral palate using the de-epithelialized gingival graft technique. After harvesting, the connective tissue graft is sutured to the recipient bed. Finally, the flap is positioned 2 mm over the cementoenamel junction and sutured with 6-0 polypropylene sutures. No periodontal dressing is applied.
  Arms: Vertically Coronally advanced flap combined with connective tissue graft
Procedure: Free gingival graft — A partial-thickness flap is elevated (using a blade #15c) with horizontal incisions at the cemento-enamel junction (CEJ) level of the adjacent teeth. Then, two vertical incisions extending to the apical are made from the two ends of the horizontal incision. The epithelium in the framed region is removed with a scalpel, and the underlying connective tissue is exposed. To achieve the best vascularization of the free gingival graft from the recipient site, bed preparation is completed with a split-thickness horizontal incision that joins the vertical incisions in the apical region. The free gingival graft is stabilized using interrupted sutures and a sling suture.
  Other Names: epithelialized free gingival graft
  Arms: Free Gingival Graft

SUMMARY:
In this comparative trial, 50 patients with shallow vestibules and Type 1/2 recessions will be treated with either a vertically coronally advanced flap + connective tissue graft or a free gingival graft. At baseline, 3rd-month, 6th-month, and 12th-month visits, the following parameters will be evaluated: buccal vestibular depth, keratinized tissue height, gingival thickness, recession depth, recession width, probing depth, and clinical attachment level. Keratinized tissue change, gingival thickness change, root coverage, clinical attachment gain, and complete root coverage will be calculated. The wound healing index, tissue appearance, patient expectations, aesthetics, and dentin hypersensitivity will be assessed at baseline and at the 6th week.

DETAILED DESCRIPTION:
Buccal vestibule depth was recorded using two different measurement methods. First, the distance between the cementoenamel junction and the deepest point of the vestibule sulcus was measured and recorded as VD1. Then, the distance between the gingival margin and the base of the vestibule sulcus was measured and recorded as VD2.

ELIGIBILITY:
Inclusion Criteria:

* full-mouth plaque and bleeding scores <15%
* the presence of at least one recession type-1/2 recession and at least one recession with recession depth ≥ 2 mm
* the presence of an identifiable cemento-enamel junction

Exclusion Criteria:

* Vestibule depth > 6mm
* Smoking > 10 cigarettes per day
* Any contraindications for periodontal surgery
* Unstable endodontic conditions or presence of any restoration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Vestibule depth 2 | Baseline
  The distance between the free gingival margin and the most apical point of the vestibul.
Vestibule depth 2 | 3rd month
  The distance between the free gingival margin and the most apical point of the vestibul.
Vestibule depth 2 | 6th month
  The distance between the free gingival margin and the most apical point of the vestibul.
Vestibule depth 2 | 12th month.
  The distance between the free gingival margin and the most apical point of the vestibul.
Vestibule depth 1 | Baseline
  The distance between the free semento-enamel junction and the most apical point of the vestibul.
Vestibule depth 1 | 3rd month
  The distance between the free semento enamel junction and the most apical point of the vestibul.
Vestibule depth 1 | 6th month
  The distance between the free semento-enamel junction and the most apical point of the vestibul.
Vestibule depth 1 | 12th month
  The distance between the free semento-enamel junction and the most apical point of the vestibul.

SECONDARY OUTCOMES:
Recession depth (RD) | Baseline
  Measured as the distance from the cementoenamel junction to the gingival margin
Recession depth (RD) | 6th week
  Measured as the distance from the cementoenamel junction to the gingival margin
Recession depth (RD) | 6th month.
  Measured as the distance from the cementoenamel junction to the gingival margin
Recession depth (RD) | 12th month.
  Measured as the distance from the cementoenamel junction to the gingival margin
Probing depth (PD) | Baseline
  Measures as the distance from the apical of gingival sulcus to the gingival margin.
Probing depth (PD) | 6th week
  Measures as the distance from the apical of gingival sulcus to the gingival margin.
Probing depth (PD) | 6th month
  Measures as the distance from the apical of gingival sulcus to the gingival margin.
Probing depth (PD) | 12th month.
  Measures as the distance from the apical of gingival sulcus to the gingival margin.
Clinical attachment level (CAL) | Baseline.
  measured as the distance from th tip of the probe inserted into the sulcus to de cementoenamel junction.
Clinical attachment level (CAL) | 6th week
  measured as the distance from th tip of the probe inserted into the sulcus to de cementoenamel junction.
Clinical attachment level (CAL) | 6th month
  measured as the distance from th tip of the probe inserted into the sulcus to de cementoenamel junction.
Clinical attachment level (CAL) | 12th month.
  measured as the distance from th tip of the probe inserted into the sulcus to de cementoenamel junction.
Keratinized tissue height (KTH) | Baseline.
  measured from the most apical point of the recession at the gingival margin to the mucogingival line.
Keratinized tissue height (KTH) | 6th week
  measured from the most apical point of the recession at the gingival margin to the mucogingival line.
Keratinized tissue height (KTH) | 6th month
  measured from the most apical point of the recession at the gingival margin to the mucogingival line.
Keratinized tissue height (KTH) | 12th month.
  measured from the most apical point of the recession at the gingival margin to the mucogingival line.
Gingival thickness (GT) | Baseline.
  determined 1.5 mm apical to the gingival margin, measured with the caliper accurete to the nearest 0.1 mm.
Gingival thickness (GT) | 6th week.
  determined 1.5 mm apical to the gingival margin, measured with the caliper accurete to the nearest 0.1 mm.
Gingival thickness (GT) | 6th month.
  determined 1.5 mm apical to the gingival margin, measured with the caliper accurete to the nearest 0.1 mm.
Gingival thickness (GT) | 12th month.
  determined 1.5 mm apical to the gingival margin, measured with the caliper accurete to the nearest 0.1 mm.
Wound healing index (WHI) | 2nd week
  Wound healing index (WHI) was recorded two-weeks after surgery. The wound surface was visually inspected and the soft tissue healing was defined as 'uneventful' (score 1), 'slightly disturbed' (score 2) or 'poor' (score 3) based on the presence and severity of the items including patient discomfort, erythema, edema, suppuration and flap dehiscence.
Tissue appearance (TA) | 6th week
  Tissue appearance (TA) was evaluated by asking the patients to score the consistency, contour, color match, keloid formation degree and contiguity of their treated sites at T2. The scores were collected as points, shown in parentheses, by asking the consistency as firm (1p) or spongy (0p); contour as presence (2p) or absence (0p) of knife-edged and scalloped gingival margin; color match as excellent (3p), good (2p), adequate (1p) or unsatisfactory (0p); keloid formation degree as absent (1p) or present (0p); contiguity as the presence (-1p) or absence (0p) of each perceptible incision mark.
Dentine hypersensitivity (DH) | 6th week
  Dentine hypersensitivity (DH) was evaluated with air evaporative stimulus method at baseline and T2. After placement of finger(s) for preserving the nearby teeth, the recession sites were subjected to evaporative stimulus comprised of 1-second air blast from 1 to 3 mm distance by using the air spray at 40-65 psi pressure and 19±50C. After application, the patients were requested to give a score to their DH between 0 (=no pain) and 10 (=extreme pain).
Patient expectations (PE) | 6th week
  Patient expectations (PE) were evaluated by requesting from the patients to rate their treatment results at T2, as satisfactory or not, in terms of appearance, experience and obtained root coverage.
Aesthetics (A) | 6th week
  Aesthetics (A) was evaluated by the patient at T1 by rating its level as excellent, good, fair or poor.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Parlak HM, Yilmaz BT, Durmaz MH, Toz H, Keceli HG. The effects of vertically coronally advanced flap and free gingival graft techniques on shallow vestibule: a randomized comparative prospective trial. Clin Oral Investig. 2023 Dec;27(12):7425-7436. doi: 10.1007/s00784-023-05332-4. Epub 2023 Oct 19. PMID 37855920